CLINICAL TRIAL: NCT03050125
Title: The Impact of Hypo-osmolar Drops on Contact Lens Comfort
Acronym: SAFFRON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Contact Lens Research (Other)
Collaborators: CooperVision, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Centre for Contact Lens Research, Director, Centre for Contact Lens Research, University of Waterloo
Organization: University of Waterloo (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 21907
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Contact Lens Related Dry Eye

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hypo-osmolar drop 1 (Experimental): Subject will receive regular instillations of hypo-osmolar sterile saline drops with the lowest osmolarity of the two hypo-osmolar drops.
  Interventions: Device: Hypo-osmolar drop 1
- Hypo-osmolar drop 2 (Experimental): Subject will receive regular instillations of hypo-osmolar sterile saline drops with the highest osmolarity of the two hypo-osmolar drops.
  Interventions: Device: Hypo-osmolar drop 2
- Iso-osmolar drop (Experimental): Subject will receive regular instillations of sterile iso-osmolar saline drops.
  Interventions: Device: Iso-osmolar drop

INTERVENTIONS:
Device: Hypo-osmolar drop 1 — 180 mOsmol sterile saline drops used as a contact lens rewetting drop.
  Arms: Hypo-osmolar drop 1
Device: Hypo-osmolar drop 2 — 240 mOsmol sterile saline drops used as a contact lens rewetting drop.
  Arms: Hypo-osmolar drop 2
Device: Iso-osmolar drop — 300 mOsmol sterile saline drops used as a contact lens rewetting drop.
  Arms: Iso-osmolar drop

SUMMARY:
This pilot study will investigate the impact of sterile saline drops that are formulated at hypo-osmolar levels on CL comfort in comparison to an iso-osmolar drop, in a group of symptomatic CL wearers.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age;
* Has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is willing and able to stay within the School of Optometry and Vision Science building for the duration of each Study Day;
* Currently wears daily, soft, frequent replacement lenses licensed in Canada (daily, bi-weekly or monthly disposable lenses, no extended wear, no monovision) for at least 3 days/week and 6 hours/day during the 2 months prior to enrolment;
* Is symptomatic according to the following classification:

  * Reports a difference between average and comfortable wear time with habitual lenses of at least 3 hours;
  * Fall into the symptomatic group as per Young's criteria (Appendix 4).
* Is able to remove and insert the lenses by themselves;
* Owns a wearable pair of spectacles;
* Is willing to wear the study lenses for 10 hours;
* Has visual acuity (VA) correctable to logMAR 0.20 or better in each eye;
* Shows an acceptable lens fit with their habitual lenses;

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has any known active* ocular disease and/ or infection;
* Has any ocular abnormality that would contraindicate contact lens wear;
* Has any known infection or inflammation that requires treatment or has a systemic condition that in the opinion of the investigator may affect the study measures;
* Is using any systemic or topical medications that in the option of the investigator may affect the study measures;
* Has any known sensitivity to the diagnostic pharmaceuticals and products to be used in this study;
* Is pregnant or lactating (by verbal communication) due to potential ocular physiology changes that may affect the study outcome;
* Is aphakic;
* Has undergone refractive error surgery;
* Is a member of the CCLR directly involved in the data collection. *For the purpose of this study, active ocular disease is defined as an infection or inflammation that requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered an active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Participant's Subjective Rating of Comfort (Questionnaire) | Baseline, 1.5hrs, 3hrs, 4.5hrs, 6hrs, 7.5hrs, 9hrs, End of 1 day
  Participants rated their eye comfort by subjective questionnaire (un-annotated scale, 0-100, 0=Very poor comfort, 100=Excellent comfort). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Participant's Subjective Rating of Dryness (Questionnaire) | Baseline, 1.5hrs, 3hrs, 4.5hrs, 6hrs, 7.5hrs, 9hrs, End of 1 day
  Participants rated the dryness of their eyes by subjective questionnaire (un-annotated scale, 0-100, 0=Very dry, 100=No dryness at all). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Participant's Subjective Rating of Foreign Body Sensation (Questionnaire) | Baseline, 1.5hrs, 3hrs, 4.5hrs, 6hrs, 7.5hrs, 9hrs, End of 1 day
  Participants rated the foreign body sensation of their eyes by subjective questionnaire (un-annotated scale, 0-100, 0=Intense feeling of foreign body sensation, 100=No foreign body sensation at all). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Participant's Subjective Rating of Stability of Vision (Questionnaire) | Baseline, 1.5hrs, 3hrs, 4.5hrs, 6hrs, 7.5hrs, 9hrs, End of 1 day
  Participants rated the stability of their vision by subjective questionnaire (un-annotated scale, 0-100, 0=Not stable at all/ very fluctuating, 100=Very stable). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Participant's Subjective Rating of Comfort (Questionnaire) - Likert scale | Baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of 1 day.
  Participants responded to the statement "My eyes feels comfortable" (5 possible ratings, Strongly agree, agree, undecided, disagree, strongly disagree). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Participant's Subjective Rating of Dryness (Questionnaire) - Likert scale | Baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of 1 day.
  Participants responded to the statement "My eyes feel dry" (5 possible ratings, Strongly agree, agree, undecided, disagree, strongly disagree). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Participant's Subjective Rating of Burning (Questionnaire) - Likert scale | Baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of 1 day.
  Participants responded to the statement "My eyes burn" (5 possible ratings, Strongly agree, agree, undecided, disagree, strongly disagree). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Participant's Subjective Rating of Awareness (Questionnaire) - Likert scale | Baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of 1 day.
  Participants responded to the statement "I am aware of the lenses in my eyes" (5 possible ratings, Strongly agree, agree, undecided, disagree, strongly disagree). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Participant's Subjective Rating of vision stability (Questionnaire) - Likert scale | Baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of 1 day.
  Participants responded to the statement "My vision is stable" (5 possible ratings, Strongly agree, agree, undecided, disagree, strongly disagree). Change over time measured at baseline, 1.5 hrs, 3 hrs, 4.5 hrs, 6 hrs, 7.5 hrs, 9 hrs and End of day.
Drop preference (compared with last drop used) | End of day 2, End of day 3
  Participant's subjective response for drop preference (compared with last drop used) at the end of days 2 and 3. (5 possible ratings: Strongly prefer Day 1, Prefer Day 1, No preference, Prefer Day 2, Strongly prefer day 2 OR Strongly Prefer Day 2, Prefer Day 2, No preference, Prefer Day 3, Strongly prefer day 3)

SECONDARY OUTCOMES:
Tear film osmolarity | Baseline, End of 1 day
  Tear film osmolarity in mOsmol/L, measured prior to the first drop of the day and at the end of the day.
Tear meniscus height | Baseline, End of 1 day
  Tear meniscus height in mm, measured prior to the first drop of the day and at the end of the day.
Non-invasive tear film break-up time (NITBUT) | Baseline, End of 1 day
  Measurement of time taken in seconds for a dry spot to appear on the corneal surface after blinking.
Conjunctival hyperemia | Baseline, 4.5 hrs, End of 1 Day
  Conjunctival hyperemia evaluated on a scale from 0 (negligible) to 100 (severe).
Limbal hyperemia | Baseline, 4.5 hrs, End of 1 Day
  Limbal hyperemia evaluated on a scale from 0 (normal) to 4 (severe).
Average corneal staining | Baseline, 4.5 hrs, End of 1 Day
  Average corneal staining evaluated on a scale from 0 (normal) to 4 (severe).
Lens movement | Baseline, 4.5 hrs, End of 1 Day
  Amount of lens movement on blink (mm).
Lens lag | Baseline, 4.5 hrs, End of 1 Day
  Amount of lens lag on blink (mm).
Lens Tightness | Baseline, 4.5 hrs, End of 1 Day
  Amount of lens tightness (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No